CLINICAL TRIAL: NCT05730712
Title: Phase II Trial of Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf (HP) Plus Enzalutamide for the Treatment of Selected Patients With Metastatic Castration-Resistant Prostate Cancer (TraPPer)
Brief Title: Pertuzumab, Trastuzumab, Hyaluronidase-zzxf and Enzalutamide for Treatment of Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210504; NCI-2022-10773 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC210504 (Other: Mayo Clinic in Rochester); 21-013057 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Castration-Resistant Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Specimen Handling; enzalutamide; Trastuzumab; pertuzumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (HP, enzalutamide) (Experimental): Patients receive pertuzumab, trastuzumab, and hyaluronidase-zzxf SC on day 1 of each cycle and enzalutamide PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO, biopsy, CT, and MRI scans and collection of blood samples throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography; Drug: Enzalutamide; Drug: Hyaluronidase-zzxf/Pertuzumab/Trastuzumab; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Drug: Hyaluronidase-zzxf/Pertuzumab/Trastuzumab — Given SC
  Other Names: Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; Pertuzumab/Trastuzumab/Hyaluronidase-zzxf; Phesgo
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well pertuzumab, trastuzumab, hyaluronidase-zzxf and enzalutamide works in treating patients with castration-resistant prostate cancer that has spread from where it first started to other places in the body (metastatic). Pertuzumab and trastuzumab are monoclonal antibodies and forms of targeted therapy that attach to a receptor protein called human epidermal growth factor receptor-2 (HER2). HER2 is found on some cancer cells. When pertuzumab or trastuzumab attach to HER2, the signals that tell the cells to grow are blocked and the tumor cell may be marked for destruction by the body's immune system. Hyaluronidase is an endoglycosidase. It helps to keep pertuzumab and trastuzumab in the body longer, so that these medications will have a greater effect. Hyaluronidase also allows pertuzumab and trastuzumab to be given by injection under the skin and shortens their administration time compared to pertuzumab or trastuzumab alone. Chemotherapy drugs, such as enzalutamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pertuzumab, trastuzumab, hyaluronidase-zzxf and enzalutamide may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the preliminary efficacy of the combination of pertuzumab, trastuzumab, and hyaluronidase-zzxf plus enzalutamide with regard to objective response rate (Prostate Cancer Clinical Trials Working Group 3 [PCWG 3.0]) in enzalutamide-refractory metastatic castration-resistant prostate cancer.

SECONDARY OBJECTIVES:

I. Estimate the radiographic progression-free survival for this combination. II. Estimate the overall survival for this combination.

EXPLORATORY OBJECTIVES:

I. Assessment of this combination for adverse events according to clinical judgment and patient-reported outcomes (Patient Reported Outcomes-Common Terminology Criteria for Adverse Events [PRO-CTCAE] - Prostate Cancer).

II. Assessment of patient quality of life using Functional Assessment of Cancer Therapy- Prostate (FACT-P) questionnaire.

CORRELATIVE OBJECTIVES:

I. Determine the correlation between outcomes as above and systemic NRG-1 levels at baseline and over time.

II. Determine the correlation between outcomes as above and change in HER2/HER3/androgen receptor (AR) gene signatures.

OUTLINE:

Patients receive pertuzumab, trastuzumab, and hyaluronidase-zzxf subcutaneously (SC) on day 1 of each cycle and enzalutamide orally (PO) once daily (QD) on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO), biopsy, computed tomography (CT), and magnetic resonance imaging (MRI) scans and collection of blood samples throughout the study.

After completion of study treatment, patients are followed up every 3 months until progressive disease then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION: Age >= 18 years.
* PRE-REGISTRATION: Clinically or histologically confirmed diagnosis of second-generation antiandrogen-refractory metastatic castration-resistant prostate cancer.
* PRE-REGISTRATION: Measurable disease as defined by the Prostate Cancer Working Group (PCWG3) criteria.
* PRE-REGISTRATION: Prior treatment required:

  * Second generation anti-androgen (2GAA) therapy (e.g., enzalutamide, abiraterone) at any time prior registration.
* PRE-REGISTRATION: Provide written informed consent.
* PRE-REGISTRATION: Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
* PRE-REGISTRATION: Ability to complete questionnaire(s) by themselves or with assistance.
* PRE-REGISTRATION: Willingness to provide mandatory blood specimens for correlative research.
* PRE-REGISTRATION: Willingness to provide mandatory tissue specimens for correlative research.
* REGISTRATION: Plasma NRG-1 level >= 4 ng/ml
* REGISTRATION: Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2.
* REGISTRATION: Hemoglobin >= 9.0 g/dL
* REGISTRATION: Absolute neutrophil count (ANC) >= 1500/mm^3
* REGISTRATION: Platelet count >= 100,000/mm^3
* REGISTRATION: Total bilirubin =< 1.5 x upper limit of normal (ULN)
* REGISTRATION: Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement).
* REGISTRATION: PT/INR/aPTT =<1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy.
* REGISTRATION: Calculated creatinine clearance >= 45 ml/min using the Cockcroft-Gault formula.
* REGISTRATION: Left ventricular ejection fraction (LVEF) >= 50% =< 15 days prior to registration.
* REGISTRATION: Provide written informed consent.
* REGISTRATION: Ability to complete questionnaire(s) by themselves or with assistance.
* REGISTRATION: Willingness to provide mandatory blood specimens for correlative research.
* REGISTRATION: Willingness to provide mandatory tissue specimens for correlative research.
* REGISTRATION: Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).

Exclusion Criteria:

* PRE-REGISTRATION: History of myocardial infarction =< 6 months prior to pre-registration, or congestive heart failure requiring use of ongoing maintenance therapy for life threatening ventricular arrhythmias.
* PRE-REGISTRATION: Failure to recover from acute, reversible effects of prior therapy regardless of interval since last treatment.

  * EXCEPTION: Grade 1 peripheral (sensory) neuropathy that has been stable for at least 3 months since completion of prior treatment.
* PRE-REGISTRATION: Uncontrolled intercurrent non-cardiac illness including, but not limited to:

  * Ongoing or active infection
  * Psychiatric illness/social situations
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
  * Any other conditions that would limit compliance with study requirements
* PRE-REGISTRATION: Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy.

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.
* PRE-REGISTRATION: Receiving any other investigational agent which would be considered as a treatment for the prostate cancer.
* PRE-REGISTRATION: Thromboembolic event =< 60 days prior to pre-registration.
* PRE-REGISTRATION: Serious cardiac illness or medical conditions including, but not confined to, the following:

  * History of NCI CTCAE v5.0 Grade >= 3 symptomatic congestive heart failure (CHF) or New York Heart Association (NYHA) Class >= II
  * High-risk uncontrolled arrhythmias (i.e., atrial tachycardia with a heart rate >= 100/min at rest, significant ventricular arrhythmia [ventricular tachycardia], or higher-grade atrioventricular [AV]-block, such as second-degree AVblock Type 2 [Mobitz II] or third-degree AV-block)
  * Serious cardiac arrhythmia or severe conduction abnormality not controlled by adequate medication
  * Angina pectoris requiring anti-angina medication
  * Clinically significant valvular heart disease
  * Evidence of transmural infarction on electrocardiogram (ECG)
  * Poorly controlled hypertension (e.g., systolic > 180 mm Hg or diastolic > 100mmHg)
* PRE-REGISTRATION: Serious cardiac arrhythmia or severe conduction abnormality not controlled by adequate medication.
* PRE-REGISTRATION: Angina pectoris requiring anti-angina medication.
* PRE-REGISTRATION: Clinically significant valvular heart disease.
* PRE-REGISTRATION: Evidence of transmural infarction on electrocardiogram (ECG).
* PRE-REGISTRATION: Poorly controlled hypertension (e.g., systolic > 180 mm Hg or diastolic > 100mmHg).
* PRE-REGISTRATION: History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias, such as structural heart disease (e.g., severe left ventricular systolic dysfunction [LVSD], left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome.
* REGISTRATION: Any of the following because this study involves an agent that has known genotoxic, mutagenic, and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential or able to father a child who are unwilling to employ adequate contraception
* REGISTRATION: Failure to recover from any of the following therapies prior to registration:

  * Major surgery
  * Chemotherapy
  * Infection requiring systemic treatment
* REGISTRATION: Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* REGISTRATION: Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy.

NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.

* REGISTRATION: Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements.
* REGISTRATION: Currently receiving any other investigational agent which would be considered as a treatment for the primary neoplasm.
* REGISTRATION: Other active malignancy =< 3 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix. NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment (e.g., other hormonal therapy, chemotherapy) for their cancer.
* REGISTRATION: History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias.
* REGISTRATION: Known hypersensitivity to pertuzumab, or trastuzumab, or hyaluronidase, or to any of its excipients.
* REGISTRATION: Requirement for drugs or substances which can interfere with the actions of the study drugs (enzalutamide or pertuzumab/trastuzumab/hyaluronidase-zzxf). Consult pharmacist for review.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of patients who experience either a partial response or complete response as defined by Prostate Cancer Working Group 3 (PCWG3).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from study entry to the first of either confirmed radiographic disease progression or death from any cause, determined based on Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria.
Overall survival (OS) | Up to 2 years
  OS is defined as the time from study entry to death from any cause.
Incidence of adverse events | Up to 1 year
  The rate of patients experiencing any Grade 3 or higher adverse event deemed at least possibly related to treatment will be reported. The maximum grade for each type of adverse event by patient will also be summarized by frequencies and percentages using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Quality of life (QoL) | Up to 1 year
  Assessed using the Functional Assessment of Cancer Therapy - Prostate (FACT-P), a 39-item questionnaire that measures quality of life (QOL) in men with prostate cancer. Questions are answered on a scale of 0-4 where 0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; and 4=very much. Patient responses to the FACT-P will be summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Orme, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT05730712/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT05730712/ICF_001.pdf